CLINICAL TRIAL: NCT07018531
Title: Vertical Soft Tissue Augmentation Using the Tent-Pole Technique With Adjunctive Therapies and Its Influence on Marginal Bone Loss Around Dental Implants: A Randomized Controlled Clinical Trial
Brief Title: Vertical Soft Tissue Augmentation With Tent Pole Technique and Its Influence on Marginal Bone Loss Around Dental Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Galimplant Dental Implants (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Full Professor in Oral Medicine, Oral Surgery and Implantology, Faculty of Dental Medicine, University of Santiago de Compostela, University of Santiago de Compostela
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 412815
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Augmentation Around Dental Implants
Keywords: Dental Implants; Vertical Soft Tissue; Tent Pole Technique; Platelet-Rich Fibrin; Photobiomodulation; Marginal Bone Loss
MeSH Terms: interventions — 9 alpha,11 alpha,15 alpha-trihydroxy-16-phenoxy-17,18,19,20-tetranorprosta-4,5,13-trienoic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tent pole technique (Experimental)
  Interventions: Procedure: VST augmentation with TPT
- Tent pole technique with platelet-rich fibrin (Experimental)
  Interventions: Procedure: TPT-PRF
- Tent pole technique with photobiomodulation (Experimental)
  Interventions: Procedure: TPT-PBM
- Negative control group (Experimental)
  Interventions: Procedure: Group control: implant placement without TPT

INTERVENTIONS:
Procedure: VST augmentation with TPT — For TPT group, vertical soft tissue augmentation will be performed simultaneously with implant placement using a 2 mm healing abutment. Than, to ensure tension-free primary closure, mucoperiosteal flaps will be mobilized through vertical releasing incisions. Wound closure will be achieved using horizontal mattress sutures, followed by simple interrupted sutures for optimal tissue adaptation. The healing abutment will act as a mechanical support to maintain space and prevent soft tissue collapse. This tented space is expected to allow blood to accumulate, clot, and gradually reorganize into connective tissue, thereby promoting an increase in vertical soft tissue thickness around the implant.
  After 2 months , the initial 2-mm healing abutment will be removed, and a 4 mm healing abutment will be placed by mading a small semilunar incision without touching the bone.
  Arms: Tent pole technique
Procedure: TPT-PRF — In the PRF group, the same surgical protocol as the TPT group will be followed. However, prior to wound closure, the tented space surrounding the healing abutment will be filled with PRF membranes.
  Arms: Tent pole technique with platelet-rich fibrin
Procedure: TPT-PBM — The PBM group will follow the same surgical protocol as the TPT group. In addition, this group will receive photobiomodulation therapy using red-light irradiation at a wavelength of 630 nm, applied to the occlusal site immediately after surgery and repeated after 7 days.
  Arms: Tent pole technique with photobiomodulation
Procedure: Group control: implant placement without TPT — The negative control group will consist of patients randomly selected from the recruited population, in accordance with the study's inclusion criteria. Participants in this group will not receive any intervention aimed at VST augmentation during implant placement. This will allow for a clear assessment of the effect of the TPT on VST gain and its impact on MBL. In accordance with ethical guidelines, patients in the control group will undergo VST augmentation at a second stage, prior to the initiation of the prosthetic phase.
  Arms: Negative control group

SUMMARY:
This study aims to evaluate the effectiveness of the tent pole technique in vertical peri-implant soft tissue augmentation and to assess its impact on marginal bone loss. Additionally, the adjunctive use of platelet-rich fibrin and photobiomodulation will be explored to determine their influence on the clinical outcomes of this procedure.

DETAILED DESCRIPTION:
Thin vertical soft tissues (VST) around dental implants pose a clinical challenge due to their strong association with marginal bone loss (MBL). Current evidence suggests that a minimum of 3 mm of VST height is essential to ensure peri-implant bone stability. Several techniques have been proposed to augment soft tissue thickness and reduce MBL, including connective tissue grafts, membranes, platelet-rich fibrin (PRF), and the Tent Pole Technique (TPT), which uses a 2 mm healing abutment to tent the soft tissue. This randomized controlled clinical trial aims to assess the effectiveness of the TPT when performed simultaneously with implant placement, in comparison to a non-intervention control group, for vertical soft tissue augmentation. Additionally, the study evaluates the impact of two adjunctive therapies: photobiomodulation (PBM) and PRF combined with TPT. In fact, PBM involves the application of low-level laser therapy at a wavelength of 630 nm to the occlusal site immediately after surgery and again at day 7, with the goal of enhancing cellular activity, accelerating healing, and promoting soft tissue regeneration. PRF, an autologous concentrate rich in growth factors, is used to fill the space created by the healing abutment in the TPT, further supporting tissue regeneration. The study includes four groups: TPT alone, TPT combined with PBM, TPT combined with PRF, and a control group without soft tissue intervention. The hypothesis is that TPT is effective in increasing vertical soft tissue thickness and maintaining marginal bone levels, and that its combination with either PBM or PRF may further enhance clinical outcomes both in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age. They should be legally capable of adhering to study protocols, which include maintaining proper oral hygiene, attending all scheduled follow-up visits, fully understanding the proposed surgical procedures, and signing the informed consent form.
* single edentulous sites in the premolar and/or molar region of the mandible.
* Vertical gingival thickness must be more than 1 mm and less than or equal to 2 mm.
* A minimum of 2 mm of attached gingiva should be present on both the buccal and lingual sides of the implant sites.
* Buccal bone thickness must be at least 1.5 mm.

Exclusion Criteria:

* Presence of general contraindications for dental implants or surgical interventions.
* Heavy smoking, defined as more than 10 cigarettes daily, including pipe, vape or cigar use.
* Poor oral hygiene, characterized by probing depths greater than 4 mm in adjacent teeth, and a full mouth plaque score (FMPS) or full mouth bleeding score (FMBS) exceeding 25% after the pre-treatment phase.
* Guided bone regeneration at the implant site.
* History of conditions or diseases that compromise bone metabolism (e.g. Paget's disease, osteoporosis) or current use of medications that may affect bone metabolism (e.g. bisphosphonates).
* History of cancer or prior radiotherapy or chemotherapy treatments for malignancy.
* Uncontrolled diabetes.
* Current pregnancy or breastfeeding status.
* Allergies to any products involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
vertical soft tissue height | 2 months , 4 months and 6 months
Marginal BoneLoss | 2 months, 4 months, 6 months

SECONDARY OUTCOMES:
PPD | 6 months
  Pocket probing depth
BOP | 6 months
  Bleeding on probing
PI | 6 months
  Plaque Index

CONTACTS AND LOCATIONS:
Locations (2):
- Oral Medicine, Oral Surgery and Implantology Unit (Medoralres), Faculty of Medicine and Dentistry, University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain
- Oral Health and Oral Rehabilitation Research Laboratory, LR12ES11, Faculty of Dental Medecine of Monastir, University of Monastir, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
data collected during our dental implant study will be made accessible to qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR